CLINICAL TRIAL: NCT06317207
Title: Reoperation for Ipsilateral Local Recurrence Following Prior Nephron-sparing Surgery: Innovative Surgical Insights From a High-volume Urological Center
Brief Title: Evaluation of the Safety of Reoperation for Ipsilateral Recurrent Tumors After Nephron-sparing Partial Nephrectomy
Acronym: LiangAH
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Chaozhao Liang, Clinical Professor, The First Affiliated Hospital of Anhui Medical University
Other Study IDs: PJ2024-01-44; 2019b07030004 (Other Grant/Funding Number: Anhui Provincial Central Government Guides Local Science and Technology Development Project-Anhui Clinical Research Ce)
Record Dates: First submitted 2024-03-09; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Renal Cell Carcinoma; Robotic Surgical Procedures
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group: patients who underwent reoperation for locally rRCC after pNSS

SUMMARY:
To evaluate the safety of reoperation in patients with renal tumors who have ipsilateral tumor recurrence after nephron-sparing partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ipsilateral local rRCC (any recurrence in the ipsilateral kidney and retroperitoneum)

Exclusion Criteria:

1. With distant metastasis;
2. Lacking essential sugery information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We collected the patients who underwent reoperation for locally rRCC after pNSS in our institution from 2013 to 2023.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Operation time | 1 week
  Operation time

SECONDARY OUTCOMES:
Estimated blood loss | 1 week
  Estimated blood loss

IPD SHARING:
Plan to Share IPD: No
All the information we will provide with the publication